CLINICAL TRIAL: NCT05184491
Title: Nitazoxanide and Lansoprazole Based Regimens for Managing Helicobacter Pylori in Egyptian Patients (NILE Study)
Brief Title: Nitazoxanide and Lansoprazole Based Regimens for H. Pylori Management
Acronym: NILE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Liver Institute, Egypt (Other)
Collaborators: Future pharmaceutical industries (Unknown)
Responsible Party: Principal Investigator, Gasser Ibrahim El-Azab, Professor of Hepatology and Gastroenterology, National Liver Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01013334106
Record Dates: First submitted 2021-11-13; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Helicobacter Pylori
Keywords: Helicobacter pylori; Eradication; nitazoxanide; Lansoprazole; LOAD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Naïve patients - ACO therapy (Active Comparator): One hundred patients naive to H. Pylori eradication therapy will receive ACO therapy for 14 days (amoxicillin 1 g with breakfast and dinner, clarithromycin 500 mg with breakfast and dinner and lansoprazole 40 mg twice daily before meals).
  Interventions: Drug: Naïve patients - ACO therapy
- Naïve patients - LNDL therapy (Experimental): One hundred patients naive to H. Pylori eradication therapy will receive LNDL therapy for 14 days (Levofloxacin 750 mg with breakfast, nitazoxanide 500 mg twice daily with meals, doxycycline 100 mg twice daily and Lansoprazole 40 mg twice daily before meals)
  Interventions: Drug: Naïve patients - LNDL therapy
- Naïve patients - MNDL therapy (Experimental): One hundred patients naive to H. Pylori eradication therapy will receive MNDL therapy for 14 days ( Moxifloxacin 400 mg with breakfast, nitazoxanide 500 mg twice daily with meals, doxycycline 100 mg twice daily and Lansoprazole 40 mg twice daily before meals)
  Interventions: Drug: Naïve patients - MNDL therapy
- Treatment-experienced patients- LNDL therapy (Experimental): One hundred patients who were unresponsive to previous eradication therapy will receive LNDL therapy for 14 days (Levofloxacin 750 mg with breakfast, nitazoxanide 500 mg twice daily with meals, doxycycline 100 mg twice daily and Lansoprazole 40 mg twice daily before meals)
  Interventions: Drug: Treatment-experienced patients- LNDL therapy
- Treatment-experienced patients- MNDL therapy (Experimental): One hundred patients who were unresponsive to previous eradication therapy will receive MNDL therapy for 14 days ( Moxifloxacin 400 mg with breakfast, nitazoxanide 500 mg twice daily with meals, doxycycline 100 mg twice daily and Lansoprazole 40 mg twice daily before meals)
  Interventions: Drug: Treatment-experienced patients- MNDL therapy

INTERVENTIONS:
Drug: Naïve patients - ACO therapy — Naïve patients will receive classic triple therapy (amoxicillin, clarithromycin and lansoprazole) for 14 days
  Arms: Naïve patients - ACO therapy
Drug: Naïve patients - LNDL therapy — Naïve patients will receive Levofloxacin, nitazoxanide, doxycycline and Lansoprazole for 14 days
  Arms: Naïve patients - LNDL therapy
Drug: Naïve patients - MNDL therapy — Naïve patients will receive Moxifloxacin, nitazoxanide, doxycycline and Lansoprazole for 14 days
  Arms: Naïve patients - MNDL therapy
Drug: Treatment-experienced patients- LNDL therapy — Experienced patients will receive Levofloxacin, nitazoxanide, doxycycline and Lansoprazole for 14 days
  Arms: Treatment-experienced patients- LNDL therapy
Drug: Treatment-experienced patients- MNDL therapy — Experienced patients will receive Moxifloxacin, nitazoxanide, doxycycline and Lansoprazole for 14 days
  Arms: Treatment-experienced patients- MNDL therapy

SUMMARY:
The study will evaluate the eradication rate and tolerability of modified LOAD regimens (three antibiotics and a proton pump inhibitor (lansoprazole)) for management of HP infection in treatment-naive patients as well as patients who failed previous therapies.

DETAILED DESCRIPTION:
This will be randomized, parallel group, comparative open-label study that will be conducted to evaluate the efficacy and tolerability of a four-drug regimen (modified LOAD regimen) in eradicating HP. The study will evaluate the efficacy of modified LOAD regimens(levofloxacin/moxifloxacin, nitazoxanide, doxycycline and lansoprazole) inpatients who failed previous therapies and compare these regimens with the classic triple therapy (amoxicillin, clarithromycin and lansoprazole) in treatment naïve patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients presented with dyspepsia for more than one month with positive H. pylori antigen test in stool

Exclusion Criteria:

* Treatment with proton pump inhibitors, bismuth, H2 receptor antagonist, or sucralfate within the two weeks before study entry, recent use of antibiotics (within one month), allergy to any of the study drugs, active bleeding, gastric surgery, pregnancy, any current malignancy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-03-15 (Estimated)

PRIMARY OUTCOMES:
Number of participants with negative results of enzyme immunoassay H. pylori antigen test in stool (Monocent, Inc., CA, USA). | 4 weeks after completion of treatment
  successful eradication of H. pylori confirmed by H. pylori antigen test in stool. Monocent, Inc.'s H. pylori Antigen Test System is an enzyme immunoassay for the qualitative and quantitative detection of H. pylori antigen in human stool. The patient has to be asked to collect the specimen avoiding any possible contact with urine or water. The patient submitted to the test should not be under antibiotic or anti-acid treatments.
  immunoassay for the qualitative and quantitative detection of H. li tiihtlIt iitdd id ithiy fthqlitti pylori antigen in human stool. diif iblHli

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by Egyptian pharmacovigilance Center (EPVC) criteria | Through study completion, an average of 24 weeks
  Safety and tolerability of these regimens will be assessed by reporting adverse events by Individual Case Safety Reports for EPVC

CONTACTS AND LOCATIONS:
Overall Officials: Gasser El-Azab, M.D., Principal Investigator — National Liver Institute
Locations (1):
- National Liver institute - Menoufia University, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: No